CLINICAL TRIAL: NCT00818454
Title: A Multicenter Randomized Study Starting With a 4 Week 2 Way Crossover Double Blind Treatment Phase Comparing the Efficacy and Safety of Combivent CFC MDI to Albuterol HFA MDI Followed by a 4 Week Open Label Combivent Respimat Treatment Phase When All Study Drugs Are Used for Symptom Relief as Needed in Pts With Moderate to Severe Asthma (GINA 2007 Treatment Steps 3-5)
Brief Title: 4 Week 2 Way Crossover Double Blind Treatment Phase With Combivent CFC Versus Albuterol Followed by a 4 Week Open Label Combivent Respimat When All Drugs Are Used for Symptom Relief as Needed in Pts With Moderate to Severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Crossover | Purpose: Treatment
Other Study IDs: 1012.57; 57948
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Results first posted 2010-11-23 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol, Ipratropium Drug Combination

INTERVENTIONS:
Drug: Combivent CFC MDI
Drug: Albuterol HFA MDI
Drug: Respimat Combivent

SUMMARY:
The primary goal of this trial is to compare the efficacy and safety of COMBIVENT CFC MDI with albuterol HFA MDI, the current standard reliever medication in asthma. In the first cross-over part of the study (Treatment Phases 1 and 2) the marketed product, COMBIVENT CFC MDI will be used. In the second, parallel group part of the trial (Treatment Phase 3) COMBIVENT RESPIMAT will be tested for acute bronchodilator efficacy in a blinded manner at the clinic visits. During the third 4-week treatment phase open label COMBIVENT RESPIMAT will be used for symptom relief as needed.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign and date an Informed Consent consistent with International Conference on Harmonization Good Clinical Practices (ICH GCP) guidelines and local regulations prior to participation in the trial (i.e., prior to any study procedures, including washout of any medication) at Visit 1.
2. Male or female patients greater to or equal to 18 years of age.
3. Physician diagnosis of moderate-to-severe asthma (GINA Guidelines) existing for >1 year.
4. Reversible airway obstruction (more than or equal to 12 % or at least 200 mL improvement in FEV1 post bronchodilator after 4 puffs of albuterol HFA MDI).
5. Pre-bronchodilator clinic measured FEV1 ≤80% of predicted normal value (measured greater to or equal to 6 hours of the last use of short acting bronchodilator and greater to or equal to 12 hours after the last use of LABA if applicable).
6. Continuous treatment with inhaled corticosteroids (ICS) with or without long-acting beta agonists (LABA) and other controller medication(s) for at least 6 weeks prior to screening (GINA 2007 Treatment Steps 3 to 5).
7. No change in dos or regimen of ICS and LABA or other controller medications (including oral corticosteroids [OCS] if applicable), for at least 2 weeks prior to Visit 2.
8. Use of short acting bronchodilator at least three times a week for symptom relief in the 2 weeks prior to Visit 1.
9. Score of ≥1.5 points on the Asthma Control Questionnaire (ACQ) (see Appendix 10.6).
10. Able to perform technically acceptable pulmonary function tests at the clinic and peak flow measurements with the eDiary/Peak Expiratory Flow Meter.
11. Able to perform all necessary recordings (symptoms and as needed medication use) in the electronic diary, which is a part of the eDiary/Peak Expiratory Flow Meter.
12. Investigator assessment of patients ability to inhale medication from a metered dose inhaler and RESPIMAT inhaler.

Exclusion Criteria:

1. Significant disease other than asthma not limited to diagnosis of COPD, such as, active tuberculosis, cystic fibrosis, alpha 1 antitrypsin deficiency, clinically significant bronchiectasis, interstitial lung disease, allergic bronchopulmonary aspergillosis, or constrictive bronchiolitis. A significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the study, or (ii) influence the results of the study, or (iii) cause concern regarding the patient ability to participate in the study.
2. History of thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion 1.
3. History of life-threatening asthma attack.
4. Worsening of asthma that required treatment with an addition or increase in OCS dose (steroid burst) in the 4- week period prior to Visit 2.
5. Current or ex-smokers who quit <1 year before enrollment. Ex-smokers who quit less than 1 year from enrollment must have a cigarette smoking history of less than 10 pack years.

   Pack years = Number of cigarettes/day x years of smoking 20
6. Use of oral beta-adrenergic agents within 4 weeks prior to screening.
7. Treatment with inhaled ipratropium, ipratropium/albuterol combination, or nasal ipratropium within 1week of Visit 2.
8. Treatment with inhaled tiotropium within 4 weeks of Visit 2.
9. Known hypersensitivity to anticholinergic drugs, benzalkonium chloride (BAC), ethylenediaminetetracetic acid (EDTA) or any other components of the tiotropium inhalation solution or MDI.
10. Known narrow-angle glaucoma.
11. Clinically relevant abnormal hematology or blood chemistry at screening if the abnormality defines a significant disease as defined in exclusion criterion 1.
12. Recent history (i.e., one year less) of myocardial infarction. Cardiac arrhythmias, newly diagnosed arrhythmias and/or any arrhythmia requiring an intervention (i.e., hospitalization, cardio version, pacemaker placement, and automatic implantable cardiac defibrillator placement) or a change in drug therapy during the last year.
13. Hospitalization for cardiac failure during the past year.
14. Malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years, with the exception of treated basal cell carcinoma.
15. Unwillingness or inability to use a highly effective method of birth control by women of childbearing potential. Highly effective methods of birth control are defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomised partner. Barrier methods of contraception are accepted if condom or occlusive cap is used together with spermicides (e.g., foam or gel). Female patients will be considered to be of childbearing potential unless surgically sterilized by hysterectomy or bilateral tubal ligation/salpingectomy, or post-menopausal for at least two years.
16. Pregnancy or nursing.
17. Any investigational drug taken within 30 days or six half-lives (whichever is greater) prior to Visit 2.
18. Previous randomization in this study or current participation in another study.
19. Symptomatic prostate hypertrophy or bladder neck obstruction. Patients with symptomatically controlled prostate hypertrophy on medications may be included and should continue their medications.
20. Use of monoamine oxidase inhibitors or tricyclic antidepressants. Examples include but are not limited to the following for monoamine oxidase inhibitors nardil, parnate, marplan and for tricyclic antidepressants: amitriptyline, norpramine, and pamelor.
21. History of and/or active alcohol or drug abuse.
22. Patient who have been treated with beta-blocker medication during the screening of the study. Topical cardio-selective beta-blocker eye medications for treatment of acute angle glaucoma are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (41):
- United States (41):
  - 1012.57.121 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1012.57.144 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1012.57.145 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1012.57.124 Boehringer Ingelheim Investigational Site, Palmdale, California
  - 1012.57.137 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1012.57.130 Boehringer Ingelheim Investigational Site, Stockton, California
  - 1012.57.134 Boehringer Ingelheim Investigational Site, Centennial, Colorado
  - 1012.57.151 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1012.57.119 Boehringer Ingelheim Investigational Site, Panama City, Florida
  - 1012.57.149 Boehringer Ingelheim Investigational Site, Winter Park, Florida
  - 1012.57.104 Boehringer Ingelheim Investigational Site, Augusta, Georgia
  - 1012.57.107 Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - 1012.57.127 Boehringer Ingelheim Investigational Site, Normal, Illinois
  - 1012.57.140 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1012.57.143 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1012.57.126 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1012.57.147 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1012.57.113 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1012.57.131 Boehringer Ingelheim Investigational Site, Plymouth, Minnesota
  - 1012.57.116 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1012.57.146 Boehringer Ingelheim Investigational Site, Bozeman, Montana
  - 1012.57.132 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1012.57.139 Boehringer Ingelheim Investigational Site, Skillman, New Jersey
  - 1012.57.109 Boehringer Ingelheim Investigational Site, Chapel Hill, North Carolina
  - 1012.57.118 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 1012.57.128 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1012.57.102 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1012.57.129 Boehringer Ingelheim Investigational Site, Lake Oswego, Oregon
  - 1012.57.138 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1012.57.108 Boehringer Ingelheim Investigational Site, Hershey, Pennsylvania
  - 1012.57.114 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1012.57.111 Boehringer Ingelheim Investigational Site, Upland, Pennsylvania
  - 1012.57.142 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 1012.57.117 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1012.57.103 Boehringer Ingelheim Investigational Site, Union, South Carolina
  - 1012.57.136 Boehringer Ingelheim Investigational Site, El Paso, Texas
  - 1012.57.148 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1012.57.101 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1012.57.141 Boehringer Ingelheim Investigational Site, Seattle, Washington
  - 1012.57.150 Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - 1012.57.105 Boehringer Ingelheim Investigational Site, Madison, Wisconsin

REFERENCES:
- [Derived] Donohue JF, Wise R, Busse WW, Garfinkel S, Zubek VB, Ghafouri M, Manuel RC, Schlenker-Herceg R, Bleecker ER. Efficacy and safety of ipratropium bromide/albuterol compared with albuterol in patients with moderate-to-severe asthma: a randomized controlled trial. BMC Pulm Med. 2016 Apr 30;16(1):65. doi: 10.1186/s12890-016-0223-3. PMID 27130202

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * Crossover Part of the Study (Treatment Period 1)
  * Crossover Part of the Study (Washout Period of 1 Week)
  * Crossover Part of the Study (Treatment Period 2)
  * Parallel Part of the Study Following Second Randomization (Treatment Period 3)
Groups:
- Albuterol HFA First, Then Combivent CFC: Albuterol Hydrofluoroalkene, Combivent Chlorofluorocarbon
- Combivent CFC First, Then Albuterol HFA: Combivent Chlorofluorocarbon, Albuterol Hydrofluoroalkene
- Placebo Respimat: Placebo Respimat (matching Combivent Respimat)
- Combivent Respimat: Combivent Respimat (contains the effective dose of albuterol)
Period: Treatment Period 1
Arm/Group | Albuterol HFA First, Then Combivent CFC | Combivent CFC First, Then Albuterol HFA | Placebo Respimat | Combivent Respimat
Started | 115 | 111 | 0 | 0
Completed | 112 | 110 | 0 | 0
Not Completed | 3 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Other | 3 | 0 | 0 | 0
Period: Washout Period of 1 Week
Arm/Group | Albuterol HFA First, Then Combivent CFC | Combivent CFC First, Then Albuterol HFA | Placebo Respimat | Combivent Respimat
Started | 112 | 110 | 0 | 0
Completed | 108 | 107 | 0 | 0
Not Completed | 4 | 3 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0
Not completed — Other | 1 | 2 | 0 | 0
Period: Treatment Period 2
Arm/Group | Albuterol HFA First, Then Combivent CFC | Combivent CFC First, Then Albuterol HFA | Placebo Respimat | Combivent Respimat
Started | 108 | 107 | 0 | 0
Completed | 106 | 106 | 0 | 0
Not Completed | 2 | 1 | 0 | 0
Not completed — Other | 2 | 1 | 0 | 0
Period: Treatment Period 3
Arm/Group | Albuterol HFA First, Then Combivent CFC | Combivent CFC First, Then Albuterol HFA | Placebo Respimat | Combivent Respimat
Started | 0 | 0 | 26 | 139
Completed | 0 | 0 | 26 | 138
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Participants randomized to crossover part at randomization 1
Arm/Group | Entire Study Population
Number analyzed (Participants) | 226
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.1 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130
  Male | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 215
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Amer. Ind./Alaska Nat | 1
  Asian | 2
  Black/African Amer. | 44
  Hawaiian/Pacif. Isle | 5
  White | 174
Body mass index [Mean (Standard Deviation); unit: Kilograms per square meter] | 31.1 (6.7)
Smoking history [Number; unit: Participants]
  Never smoked | 163
  Ex-smoker | 63
  Currently smokes | 0
Alcohol history [Number; unit: Participants]
  Non drinker | 76
  Drinks - no interference | 150
  Drinks - possible interference | 0
Height [Mean (Standard Deviation); unit: Centimeters] | 169.9 (11.0)
Weight [Mean (Standard Deviation); unit: Kilograms] | 89.9 (21.0)

OUTCOME MEASURES:

1. Primary Outcome: FEV1 AUC0-6 Response (Crossover Part of the Study)
Description: Change from baseline after 4 weeks in Forced Expiratory Volume Area Under (FEV1 AUC) the Curve from 0 to 6 hours.
Time Frame: Test day baseline and test day FEV1 AUC 0-6, after 4 weeks
Population: Full analysis set 1 (FAS1) consisted of all patients who were dispensed study medication, were documented to have taken at least one dose of investigational treatment, and had non-missing Visit 3 baseline values and non-missing responses for both peak FEV1 and FEV1 AUC0-6 at Visit 3.
Measure: Least Squares Mean (Standard Error); unit: liters
Groups:
- Albuterol HFA: Albuterol Hydrofluoroalkene
- Combivent CFC: Combivent Chlorofluorocarbon
Arm/Group | Albuterol HFA | Combivent CFC
Number analyzed (Participants) | 191 | 193
liters | 0.167 (0.026) | 0.252 (0.026)
Statistical Analysis 1: Comparison: Albuterol HFA vs Combivent CFC; Test type: Superiority or Other; p < 0.0001, MMRM ANCOVA

2. Primary Outcome: Peak FEV1 Response (Crossover Part of the Study)
Description: Change from baseline after 4 weeks in peak Forced Expiratory Volume response
Time Frame: Test day baseline and test day peak FEV1, after 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Albuterol HFA | Combivent CFC
Number analyzed (Participants) | 191 | 193
liters | 0.357 (0.031) | 0.434 (0.031)
Statistical Analysis 1: Comparison: Albuterol HFA vs Combivent CFC; Test type: Superiority or Other; p < 0.0001, MMRM ANCOVA

3. Secondary Outcome: Mini Asthma Quality of Life Questionnaire (Crossover Part of the Study)
Description: Change from baseline after 4 weeks in Mini-AQLQ score. Worst score - 1 (most severe), best score - 7 (less severe)
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Albuterol HFA | Combivent CFC
Number analyzed (Participants) | 191 | 193
Scores on scale | 0.150 (0.05) | 0.220 (0.05)
Statistical Analysis 1: Comparison: Albuterol HFA vs Combivent CFC; Test type: Superiority or Other; p = 0.159, MMRM ANCOVA

4. Secondary Outcome: Asthma Control Questionnaire (Crossover Part of the Study)
Description: Change from baseline after 4 weeks in ACQ score. Worst score - 6(most severe), best score - 0 (no symptoms)
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Albuterol HFA | Combivent CFC
Number analyzed (Participants) | 191 | 193
Scores on scale | -0.25 (0.04) | -0.25 (0.04)
Statistical Analysis 1: Comparison: Albuterol HFA vs Combivent CFC; Test type: Superiority or Other; p = 0.8278, MMRM ANCOVA

5. Secondary Outcome: Puffs Study Medication Used During Day (Crossover Part of the Study)
Description: Change from baseline in weekly mean of puffs of blinded study medication (albuterol HFA or combivent CFC) used during day
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs
Arm/Group | Albuterol HFA | Combivent CFC
Number analyzed (Participants) | 176 | 178
Puffs | -0.49 (0.07) | -0.53 (0.07)
Statistical Analysis 1: Comparison: Albuterol HFA vs Combivent CFC; Test type: Superiority or Other; p = 0.5098, MMRM ANCOVA

6. Secondary Outcome: Puffs Study Medication Used During Night (Crossover Part of the Study)
Description: Change from baseline in weekly mean of puffs of blinded study medication (albuterol HFA or combivent CFC) used during night
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs
Arm/Group | Albuterol HFA | Combivent CFC
Number analyzed (Participants) | 178 | 180
Puffs | -0.10 (0.05) | -0.12 (0.05)
Statistical Analysis 1: Comparison: Albuterol HFA vs Combivent CFC; Test type: Superiority or Other; p = 0.6591, MMRM ANCOVA

7. Secondary Outcome: Puffs Open-label Albuterol Used During Day (Crossover Part of the Study)
Description: Change from baseline in weekly mean of puffs of open-label albuterol used during day
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs
Arm/Group | Albuterol HFA | Combivent CFC
Number analyzed (Participants) | 176 | 178
Puffs | -2.24 (0.05) | -2.28 (0.05)
Statistical Analysis 1: Comparison: Albuterol HFA vs Combivent CFC; Test type: Superiority or Other; p = 0.3631, MMRM ANCOVA

8. Secondary Outcome: Puffs Open-label Albuterol Used During Night (Crossover Part of the Study)
Description: Change from baseline in weekly mean of puffs of open-label albuterol used during night
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs
Arm/Group | Albuterol HFA | Combivent CFC
Number analyzed (Participants) | 178 | 180
Puffs | -0.92 (0.02) | -0.93 (0.02)
Statistical Analysis 1: Comparison: Albuterol HFA vs Combivent CFC; Test type: Non-Inferiority or Equivalence — Enter additional comments here, if non-inferiority or equivalence analysis; p = 0.6787, MMRM ANCOVA

9. Secondary Outcome: FEV1 AUC0-6 Response (Parallel Part of the Study)
Description: Change from baseline after 4 weeks in Forced Expiratory Volume Area Under the Curve from 0 to 6 hours
Time Frame: Test day baseline and test day FEV1 AUC 0-6, after 4 weeks
Population: These analyses were done on FAS2. FAS2 is all patients who were dispensed study medication, were documented to have taken at least one dose of investigational treatment, and had a non-missing Visit 7 baseline value and non-missing responses for both peak FEV1 and FEV1 AUC0-6 at Visit 7.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo Respimat | Combivent Respimat
Number analyzed (Participants) | 26 | 139
liters | 0.041 (0.046) | 0.236 (0.020)
Statistical Analysis 1: Comparison: Placebo Respimat vs Combivent Respimat; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Adjusted for baseline, period, week, and treatment by week interaction

10. Secondary Outcome: Peak FEV1 Response
Description: Change from baseline after 4 weeks in peak Forced Expiratory Volume response
Time Frame: Test day baseline and test day peak FEV1, after 4 weeks
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo Respimat | Combivent Respimat
Number analyzed (Participants) | 26 | 139
liters | 0.199 (0.053) | 0.412 (0.023)
Statistical Analysis 1: Comparison: Placebo Respimat vs Combivent Respimat; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Adjusted for baseline, period, week, and treatment by week interaction

ADVERSE EVENTS:
Time Frame: 29 days (Treatment phase 1) + 29 days (Treatment phase 2) + 29 days (Treatment phase 3)
Arm/Group | Albuterol HFA First, Then Combivent CFC | Combivent CFC First, Then Albuterol HFA | Placebo Respimat | Combivent Respimat
Serious Adverse Events (participants affected / at risk) | 1/222 | 1/219 | 0/26 | 0/139
Other Adverse Events (participants affected / at risk) | 1/222 | 11/219 | 0/26 | 0/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albuterol HFA First, Then Combivent CFC (N=222) | Combivent CFC First, Then Albuterol HFA (N=219) | Placebo Respimat (N=26) | Combivent Respimat (N=139)
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Albuterol HFA First, Then Combivent CFC (N=222) | Combivent CFC First, Then Albuterol HFA (N=219) | Placebo Respimat (N=26) | Combivent Respimat (N=139)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 11 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.